CLINICAL TRIAL: NCT05641116
Title: Effectiveness of an Intervention Combining Adapted Physical Activity and Therapeutic Education in Patients With Chronic Symptoms Attributed to Lyme Borreliosis. Multicenter, Controlled, Randomized Pilot Study
Brief Title: Effectiveness of an Intervention Combining Adapted Physical Activity and Therapeutic Education in Patients With Chronic Symptoms Attributed to Lyme Borreliosis.
Acronym: LyMouv'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22CH398; 2022-A01120-43 (Other: ANSM)
Record Dates: First submitted 2022-11-08; First posted 2022-12-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Lyme Borreliosis; Physical Activity; Lyme Borreliosis, Nervous System
Keywords: sedentary time; therapeutic education of the patient; adapted physical activity; training program
MeSH Terms: conditions — Lyme Disease; Motor Activity; Lyme Neuroborreliosis; Sedentary Behavior | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyme Borreliosis with physical activity program (Experimental): Referral of the patient to the sport-health center of his department by the investigating physician (in connection with the attending physician for the prescription of Adaptive Physical Activity): for 24 sessions of APA for 3 months at a rate of 2 sessions/week at the sport and health center + 9 sessions of Therapeutic Patient Education in telecare
  Interventions: Other: physical activity program
- Lyme Borreliosis patients with physical activity at home (Other): routine clinical practice : encouragement by the attending physician to modify lifestyle habits with advice on resuming regular physical activity independently and combating sedentariness. At home, in autonomy for 3 months.
  Interventions: Other: Advice and recommendations of physical activity at home

INTERVENTIONS:
Other: physical activity program — 24 face-to-face APA sessions at the sport and health center for 3 months at a rate of 2 sessions per week near his home and 9 therapeutic patient education workshops for 3 months at a rate of 3 workshops per month (telecare).
  Arms: Lyme Borreliosis with physical activity program
Other: Advice and recommendations of physical activity at home — Advice and recommendations of physical activity at home (= current clinical practice in autonomy for 3 months).
  Arms: Lyme Borreliosis patients with physical activity at home

SUMMARY:
Lyme borreliosis, commonly known as Lyme disease, has been clinically described for more than a century, but has been officially recognized for 40 years, with the detection of the Borrelia bacterium by W. Burgdorfer, in ticks of the Ixodes ricinus complex, identified a few years before.

DETAILED DESCRIPTION:
Apart from the early localized presentation, with a well established treatment, Lyme borreliosis is a complex infection. Indeed, its presentation can be late and very polymorphic, which can evoke functional somatic disorders and make its management difficult. In 2016, the French Ministry of Health decided to launch a national plan to fight Lyme borreliosis. One of the objectives of this national plan was to improve management based on a specific multidisciplinary care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to the reference center for tick-borne diseases by his attending physician
* Duration of symptoms >6 months
* At the end of the initial assessment, the diagnosis of functional somatic disorders is retained after consensus between the physicians
* Patient practicing less than 150 minutes of regular physical activity per week (WHO recommendations)

Exclusion Criteria:

* Patients with cardiac or respiratory pathologies that contraindicate the practice of physical activity physical activity
* Important comorbidities contraindicating the practice of physical activity: associated cardiac pathologies associated cardiac pathologies (severe rhythm disorders such as rapid atrial fibrillation), respiratory pathologies respiratory pathologies (obstructive or severe restrictive respiratory insufficiency), disabling joint pathologies joint pathologies (gonarthrosis or coxarthrosis limiting training on a treadmill or on a high-intensity bicycle). intensity cycling).
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Average level of moderate to vigorous physical activity (PA) - MET-h/week | 1 year after implementation of the PA program
  MET = metabolic equivalent
  This is measured with actimetry (Actigraph GT3x, Pensacola, Florida, USA).

SECONDARY OUTCOMES:
average level of sedentary lifestyle (h/day) | at Month 3, Month 6 and Month 12 after implementation of the PA program
  This is measured with actimetry (Actigraph GT3x, Pensacola, Florida, USA).
  The average sedentary time measured in industrialized countries is about 4 hours per day (excluding time spent sitting at work and in transport)
Average level of moderate to vigorous physical activity (PA) - MET-h/week | at Month 3, Month 6 and Month 12 after implementation of the PA program
  This measured with Adult Physical Activity Questionnaire (APAQ) Score from 0 to 21 points, 0 = no difficulty, and 21= major difficulties.
Average level of sedentary lifestyle (h/day) | at Month 3, Month 6 and Month 12 after implementation of the PA program
  This measured with Adult Physical Activity Questionnaire (APAQ) Score from 0 to 21 points, 0 = no difficulty, and 21= major difficulties.
VO2max (in ml/min/kg) | at Month 3, Month 6 and Month 12 after implementation of the PA program
  This physical ability is measured with a cardiorespiratory test on a cycloergometer
Biceps muscular strength (kg) | at Month 3, Month 6 and Month 12 after implementation of the PA program
  Muscular strength will be assessed by biceps muscle strength (in kilograms) on the Handgrip (JAMAR Hand Dynamometer, UK)
Patient Global Impression of Change (PGIC) | at Month 3, Month 6 and Month 12 after implementation of the PA program
  Health status will be assessed by the Patient Global Impression of Change (PGIC) and measured on a 7-point Likert scale, rated from 1 for "much worse" to 7 for "much better".
Hospital Anxiety and Depression Scale (HADS) | at Month 3, Month 6 and Month 12 after implementation of the PA program
  Psychological distress will be assessed using the Hospital Anxiety and Depression Scale (HADS) The HADS scale has 14 items scored from 0 to 3. 7 questions concern anxiety and 7 others the depressive dimension, which makes it possible to obtain two scores (maximum score for each score = 21). A score greater than or equal to 11 means that the anxiety or depression is anxiety or depression is certain.
Number of patients involved in the intervention | at Month 6 after implementation of the PA program
  Assessment of adherence as measured by the number of patients involved in the intervention
medico-economic impact of the care organization | at Month 12 after implementation of the PA program
  Average cost saved per 100 patients treated in the "physical activity program group" compared to the "control group"

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU de Saint Etienne
Locations (2):
- France (2):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No